CLINICAL TRIAL: NCT02219425
Title: Gene Expression Analysis of the Endometrium After Endometrial Biopsy in Fertile Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Miacol-2014-2H
Record Dates: First submitted 2014-07-11; First posted 2014-08-18 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-08

CONDITIONS: Infertility
Keywords: Infertility; Endometrium; Endometrial biopsy; Gene expression
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- endometrial biopsy (Other)
  Interventions: Procedure: endometrial biopsy

INTERVENTIONS:
Procedure: endometrial biopsy
  Other Names: Pipelle de Cornier

SUMMARY:
The aim of this study is to evaluate the gene expression of the endometrium after an endometrial biopsy in fertile women using Next Generation Sequencing of total RNA.

DETAILED DESCRIPTION:
An endometrial biopsy is done at cycle day LH+7 and repeated in the next cycle at cycle day LH+7.

Tissue is analysed and compared for changes in gene expression profile using Seq RNA

ELIGIBILITY:
Inclusion Criteria:

* Fertile women
* Age: 18-40 years
* BMI: 18-32
* Regular menstrual cycle
* No use of hormonal contraceptives or IUD the last 3 months

Exclusion Criteria:

* Patients in need of a interpreter
* Suspected intrauterine abnormalities
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Gene Expression of the Endometrium after an endometrial biopsy | 1 month between each biopsy
  An endometrial biopsy is done at cycle day LH+7 and repeated in the next cycle at cycle day LH+7.
  Endometrial tissue is analysed for changes in gene expression profile of various chemokines and cytokines using RNA Sequencing technology

CONTACTS AND LOCATIONS:
Overall Officials: Axel Forman, MD, DMsc, Study Director — Departement of Gynaecology and Obstetrics, Aarhus University; Mia Steengaard Olesen, MD, Principal Investigator — Fertility Clinic Horsens Hospital, Aarhus University
Locations (1):
- Fertility Clinic Horsens Hospital, Horsens, Denmark